CLINICAL TRIAL: NCT07196072
Title: A Multi-component, Person-centered, and Yoga-based Coaching Program for Lupus Chronic Pain
Acronym: MiPAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Principal Investigator, Dominique Lynn Kinnett-Hopkins, Research Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00264850
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: SLE (Systemic Lupus); Chronic Pain
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a single site, single-arm, and open label feasibility study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MiPAL participant (Experimental): All study participants who meet eligibility criteria.
  Interventions: Behavioral: MiPAL

INTERVENTIONS:
Behavioral: MiPAL — MiPAL participants meet with a coach to co-develop a self-directed yoga practice based on individual preferences and limitations.

SUMMARY:
This research will assess the feasibility of a tailored yoga coaching program for reducing pain-related symptoms among people with systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and speak English sufficiently to allow for informed consent and active participation in the intervention sessions.
2. Diagnosed with systemic lupus erythematosus (SLE). In this study, SLE is classified as meeting the 2019 European League Against Rheumatism/American College of Radiology (ACR) criteria for SLE.
3. Stable doses of lupus-related medications, including prednisone, for 3 months prior to study entry.
4. Reports pain lasting ≥ 3 months and has a sum of ≥8 on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29+2 Pain Interference items (assessed at screening).
5. Willingness to attend all study visits, including attending recorded virtual coaching sessions for the duration of study.
6. Willingness to engage in yoga practices outlined in the MiPAL program.
7. Access to necessary resources for participating in a remote intervention, including a smartphone, computer, or tablet with internet

Exclusion Criteria:

1. Taking >10 mg of prednisone (or equivalent steroid dose) per day.
2. Unable to attend study visits.
3. Pregnancy.
4. Concurrent participation in other behavioral, psychotherapeutic, or pharmacological trials.
5. Any impairment, activity, or situation that in the judgment of the study team would prevent satisfactory completion of the study protocol. For example, any condition that impairs the ability to give consent or participate fully in the study.
6. Currently engaged in or starting any therapies (physical, occupational, CBT, psychotherapy, etc.) that are focused on managing chronic pain. Participants may be withdrawn from the study if they start any such therapies during their study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants recruited | Baseline, when participants complete informed consent and enroll in the study.
  Defined by the number of participants who enroll in the study compared to the target recruitment number (i.e., n=15 anticipated)
Proportion of enrolled participants who complete the study protocol | End of participation, up to 13 weeks
  The proportion of enrolled participants who complete the study protocol (i.e., study activities for the 13-week follow up)

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) score | Up to 13 weeks
  This is a 1-item survey that measures patient perceptions of intervention success. This survey is scored from 1 to 7, where lower scores indicate a better outcome.
  Researchers will consider the intervention to make participants feel better overall if their score = 1, 2, or 3

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Kinnett-Hopkins, PhD, Principal Investigator — University of Michigan; Rachel Bergmans, MPH, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No